CLINICAL TRIAL: NCT04499742
Title: Does Rise in Breath Hydrogen During Endoscopically Assisted Glucose Breath Test (EAGBT) Correlate With Radio-Isotope Location in Small Bowel: Improving Detection of Distal SIBO
Brief Title: Comparative Assessment of Radioisotope Glucose and Breath Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, MD, PhD, Augusta University
Other Study IDs: 1328690
Record Dates: First submitted 2019-02-19; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Small Intestinal Bacterial Overgrowth
MeSH Terms: interventions — Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Breath samples will be analyzed using gas chromatography for hydrogen and methane values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: Using Isotope (Tc99m-Sulfur Colloid) to label glucose and administer this directly into duodenum. — Patients will be undergoing Standard of Care procedure EAGBT for collection of duodenal fluid (aspirate and culture) and placement of a catheter into the duodenum. This catheter will be used for infusion of glucose isotope into the small bowel. Subsequently Standard of Care nuclear medicine imaging will be used to track the location of the isotope in the gut.

SUMMARY:
This is a research study about improving our diagnostic method for small intestinal bacterial overgrowth (SIBO). Patients undergoing Standard of Care (SOC) Endoscopically assisted glucose breath test (EAGBT) will undergo upper endoscopy and glucose breath tests. In this study, investigators wish to utilize Nuclear Medicine techniques to locate where the glucose solution that is administered during EAGBT is being consumed by bacteria is in the small bowel when it detects SIBO.

DETAILED DESCRIPTION:
Small intestinal bacterial overgrowth (SIBO) is characterized by bloating, gas, distention, and diarrhea due to colonization and an excessive amount of bacteria in the small bowel. Distal SIBO is the presence of excessive amounts of bacteria in the distal jejunum and/or ileum. Diagnosis of SIBO requires either duodenal aspirate with culture analysis or more commonly with breath hydrogen/methane testing. Hydrogen breath testing often uses either oral glucose or lactulose solutions. If bacteria are present in the small bowel they will ferment glucose or lactulose, producing hydrogen or methane as a byproduct. These gases are absorbed into the bowel, and then eliminated via pulmonary expiration. By detecting a rise in breath H2 and CH4 values compared to baseline, SIBO can be diagnosed. However, after oral ingestion, the majority of the glucose substrate is absorbed in the duodenum and proximal jejunum. Therefore, Glucose breath test (GBT) is good for the detection of proximal SIBO, but misses distal SIBO.

Investigators have recently shown that glucose administration into the distal duodenum through upper endoscopy has a higher positive yield for SIBO in patients with negative oral GBT. However, it is unclear if the rise in breath H2 or CH4 is because of glucose fermentation by bacteria in the distal small bowel or from fermentation by bacteria in the colon, i.e. false-positive test. Study objective here is to administer a radio-labeled glucose solution into the duodenum via an endoscopically placed nasoduodenal tube, and then determine if the rise in breath hydrogen and/or methane correlates with the location of the isotopic glucose solution in the bowel by simultaneous nuclear imaging. Results of breath testing will also be compared with duodenal aspirate/cultures taken at the time of endoscopy. Clinical response to treatment will be assessed on follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent gas, bloating, distension, and suspected SIBO
* Negative oral GBT
* 18 years and older

Exclusion Criteria:

* Pregnancy
* Diabetes
* Previous abdominal surgery except cholecystectomy, appendectomy
* Diet prep non-adherence
* Smoking or exercise causing hyperventilation prior to exam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients exhibiting SIBO symptoms.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-12-14 (Estimated); Study Completion 2021-12-14 (Estimated)

PRIMARY OUTCOMES:
Correlation between GBT result and isotope detection in small bowel | February 6, 2019 (anticipated) - December 14, 2021 (anticipated)
  Overall correlation (positive and negative) between the location of glucose isotope in small bowel (imaging) and changes in in hydrogen and methane values obtained during the breath test.

SECONDARY OUTCOMES:
Diagnostic yield of EAGBT compared to oral GBT | February 6, 2019 (anticipated) - December 14, 2021 (anticipated)
  We will compare the yield (positive, negative and overall) of endoscopic assisted GBT versus orally administered GBT
Diagnostic yield of EAGBT compared to duodenal aspirate and culture | February 6, 2019 (anticipated) - December 14, 2021 (anticipated)
  We will compare the positive and negative yield of EAGBT with the positive (>1000 CFU/ml) or negative yield of aerobic and anaerobic cultures.
Symptom patterns and demographics | February 6, 2019 (anticipated) - December 14, 2021 (anticipated)
  Compare the gas and bloating symptom patterns, clinical characteristics predisposing factors including underlying dysmotility and other demographic features between patients with positive and negative EAGBT and cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University Digestive Health Research, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No